CLINICAL TRIAL: NCT04240171
Title: Comparative Study of Dapagliflozin Versus Glimepiride Effect on Insulin Regulated Aminopeptidase (IRAP) and Interleukin-34 (IL-34) in Patient With Type 2 Diabetes Mellitus
Brief Title: Dapagliflozin Versus Glimepiride Effect in Patient With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Clinical Pharmacy Lecturer, Damanhour University
Other Study IDs: Dapagliflozin in T2DM
Record Dates: First submitted 2019-09-15; First posted 2020-01-27 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; glimepiride

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dapagliflozin: Group 1(n=30): are the patients who are prescribed dapagliflozin to control their blood sugar level.
  Interventions: Drug: Dapagliflozin 5Mg Tab
- glimepiride: Group 2 (n=30): are the patients who are prescribed glimepiride
  Interventions: Drug: Glimepiride 4Mg Tab

INTERVENTIONS:
Drug: Dapagliflozin 5Mg Tab — Dapagliflozin 5mg tablets daily
  Other Names: Diglifloz
  Groups: dapagliflozin
Drug: Glimepiride 4Mg Tab — Glimepiride Tablets daily
  Other Names: Amaryl
  Groups: glimepiride

SUMMARY:
Research objectives:

The aim of the study to check the effect of Dapagliflozin versus Glimepiride on insulin regulated aminopeptidase (IRAPe), NT-Pro BNP and interleukin-34 (IL-34) in patients with type 2 diabetes mellitus, and associated it with insulin resistance.

DETAILED DESCRIPTION:
Method and proposal steps:

1. Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University.
2. All participant agreed to take part in this clinical study and provide informed consent.
3. 60 Patients with type 2 DM will be enrolled Internal Medicine Department, Tanta University Hospital.
4. Serum samples will be collected for measuring the biomarkers.
5. All enrolled 60 patients will be mentioned as two groups; Group 1(n=30): are the patients who are prescribed dapagliflozin to control their blood sugar level. Group 2 (n=30): are the patients who are prescribed glimepiride
6. All patients will be followed up during 3 months' period.
7. At the end of 3 months, step 4 will be repeated.
8. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
9. Measuring outcomes: the primary outcome is the change from baseline to post-treatment insulin sensitivity reflected by change of serum level of measured marker after 3 months.
10. Results, discussion, conclusion, and recommendations will be given.

Methodology:

1. Fasting blood glucose (FBG) 2 hrs. post prandial blood glucose(2hPPBG) will be measured by glucometer.
2. HbA1c %, Fasting plasma insulin (FPI), Interleukin-34 (IL-34), NT-Pro BNP and extracellular domain of insulin regulated aminopeptidase (IRAPe) will be assayed by Enzyme-Linked Immunosorbent Assay (ELISA).
3. Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. 60 Patients with type 2 DM diagnosed clinically. The age ranged from 18 to 70 years. There are no limits to the duration of DM and gender.
2. HbA1c ≥ 7

Exclusion Criteria:

1. Other types of DM
2. Hypersensitivity to the drug
3. Abnormal liver function
4. Patients with renal impairment (eGFR ≤ 60 ml/min)
5. Previous history of bladder cancer

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3- 60 Patients with type 2 DM will be enrolled Internal Medicine Department, Tanta University Hospital.
  4- Serum samples will be collected for measuring the biomarkers. All enrolled 60 patients will be mentioned as two groups; Group 1(n=30): are the patients who are prescribed dapagliflozin to control their blood sugar level. Group 2 (n=30): are the patients who are prescribed glimepiride
  * All patients will be followed up during 3 months' period.
  * At the end of 3 months, step 4 will be repeated.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Blood Sugar (mg/dl) | three months
  serum blood glucose
HbA1c % | three months
  Glycated Hemoglobin

SECONDARY OUTCOMES:
NT-Pro BNP (ng/ml) | Three Months
  Natriuretic peptide tests measure levels of BNP or NT-proBNP in the blood.
IRAPe (ng/ml) | Three Months
  extracellular part of insulin-regulated aminopeptidase (IRAPe).
IL-34 (pg./ml) | Three Months
  interleukin (IL)-34.

CONTACTS AND LOCATIONS:
Overall Officials: Nashwa EL-Gharabawy, Lecturer, Study Chair — Tanta University; Rehab Werida, Study Director — Damanhour University, Faculty of Pharmacy
Locations (1):
- Tanta University Hospital, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monami M, Nardini C, Mannucci E. Efficacy and safety of sodium glucose co-transport-2 inhibitors in type 2 diabetes: a meta-analysis of randomized clinical trials. Diabetes Obes Metab. 2014 May;16(5):457-66. doi: 10.1111/dom.12244. Epub 2013 Dec 29. PMID 24320621
- [Result] Abdul-Ghani MA, Norton L, DeFronzo RA. Renal sodium-glucose cotransporter inhibition in the management of type 2 diabetes mellitus. Am J Physiol Renal Physiol. 2015 Dec 1;309(11):F889-900. doi: 10.1152/ajprenal.00267.2015. Epub 2015 Sep 9. PMID 26354881
- [Result] Davidson JA, Kuritzky L. Sodium glucose co-transporter 2 inhibitors and their mechanism for improving glycemia in patients with type 2 diabetes. Postgrad Med. 2014 Oct;126(6):33-48. doi: 10.3810/pgm.2014.10.2819. PMID 25414933
- [Derived] Zekry R, Omran GA, El-Gharbawy NM, Werida RH. Comparative study of Dapagliflozin versus Glimepiride effect on insulin regulated aminopeptidase (IRAP) and interleukin-34 (IL-34) in patient with type 2 diabetes mellitus. Sci Rep. 2023 Apr 18;13(1):6302. doi: 10.1038/s41598-023-33417-3. PMID 37072577